CLINICAL TRIAL: NCT07119177
Title: Long-Term Effects of Gestational Diabetes Mellitus on Postpartum Chronic Non-Communicable Diseases: A Prospective Cohort Study
Brief Title: Long-term Evaluation of Gestational Endocrine & Metabolic Dynamics
Acronym: LEGEND
Status: Recruiting | Type: Observational
Sponsor: Yang ZHANG (Other)
Collaborators: National Institute of Health Data Science at Peking University (Unknown)
Responsible Party: Sponsor-Investigator, Yang ZHANG, Associated chief of the endocrinology department of peking university first hospital, Peking University First Hospital
Organization: Peking University First Hospital (Other)
Other Study IDs: GDM00120241114; 2024IR33 (Other Grant/Funding Number: Peking university first hospital)
Record Dates: First submitted 2025-06-03; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Gestational Diabetes Mellitus (GDM); Non-communicable Chronic Diseases
Keywords: Gestational Diabetes Mellitus; Long-term Impact; Non-communicable Chronic Diseases; Prospective Cohort; Predictive Model
MeSH Terms: conditions — Diabetes, Gestational; Noncommunicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Gestational diabetes mellitus (GDM) is the most common complication and metabolic disorder during pregnancy, with clear risks to both the mother and fetus. In recent years, the long-term chronic diseases and poor prognosis in GDM women after delivery, as well as the risk of obesity and metabolic disorders in their offspring, have become key research topics. However, due to the long duration of GDM's impact on both the mother and offspring and its involvement in multiple disciplines, high-quality cohort studies are scarce. As a result, there is no definitive conclusion regarding the high-risk factors, natural progression, key mediators, timing of interventions, and targets for GDM's long-term effects on mothers and their offspring. This project intends to initiate a prospective follow-up study, establish a specialized cohort for the long-term effects of GDM on both mothers and their offspring, and complete the characterization of the natural course of non-communicable chronic diseases (NCDs) in GDM women and their offspring. The study will also explore high-risk and mediator factors, and develop predictive models. The goal is to provide education, postpartum follow-up, monitoring, and possibly initiate primary prevention for GDM women to reduce the long-term NCD risks, ultimately improving their life expectancy and providing a theoretical basis for intervention.

Inclusion Criteria:

1. Adult patients (≥18 years old) who registered for antenatal care and delivered at Peking University Firest Hospital's obstetrics department between 2007 and 2016.
2. Diagnosed with gestational diabetes mellitus (GDM) during pregnancy via an oral glucose tolerance test (OGTT).
3. Signed informed consent.

Exclusion Criteria:

1. Lack of pregnancy-related obstetric follow-up records.
2. Inability to cooperate with and complete subsequent scheduled follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years old) who registered for antenatal care and delivered at Peking University Firest Hospital's obstetrics department between 2007 and 2016.
* Diagnosed with gestational diabetes mellitus (GDM) during pregnancy via an oral glucose tolerance test (OGTT).
* Signed informed consent.

Exclusion Criteria:

* Lack of pregnancy-related obstetric follow-up records.
* Inability to cooperate with and complete subsequent scheduled follow-ups.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Gestational diabetes mellitus (GDM) patients who delivered at Peking University First Hospital between 2007 and 2016 will be identified through electronic medical record searches. We intend to enroll a total of 800 GDM patients meeting the above inclusion/exclusion criteria and their offspring.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2025-03-29 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of type 2 diabetes mellitus | At 8-17 years postpartum
  Subjects who meet either criterion 1 or 2 will be considered to have type 2 diabetes：
  1. With classical symptoms of diabetes: if any one of the following is met:
     Random plasma glucose ≥ 11.1 mmol/L, or Fasting plasma glucose (FPG) ≥ 7.0 mmol/L, or 2-hour plasma glucose during an oral glucose tolerance test (OGTT) ≥ 11.1 mmol/L, or HbA1c (glycated hemoglobin) ≥ 6.5%.
  2. Without classical symptoms of diabetes: either two glucose indicators measured at the same time point reaching or exceeding diagnostic thresholds, or Glucose indicators measured at two different time points reaching or exceeding diagnostic thresholds (excluding random plasma glucose).
Prevalence of metabolic syndrome | At 8-17 years postpartum
  Individuals meeting 3 or more of the following 5 components will be considered to have metabolic syndrome:
  1. Waist circumference ≥ 85 cm in women;
  2. FPG ≥ 6.1 mmol/L and/or 2hPG ≥ 7.8 mmol/L, and/or previously diagnosed diabetes;
  3. Blood pressure ≥ 130/85 mmHg, and/or previously diagnosed hypertension and treated;
  4. Fasting TG ≥ 1.7 mmol/L;
  5. Fasting HDL-C < 1.04 mmol/L.
Prevalence of cardiovascular diseases | At 8-17 years postpartum
  The presence of any of the following items is considered indicative of cardiovascular disease:
  1. Inquire about history(definitively diagnosed by a qualified physician) of cardiovascular diseases, including coronary heart disease, hypertension and arrhythmia.
  2. Quantify coronary artery calcium score via non-contrast CT scan, > 100 indicates elevated risk for coronary heart disease.
  3. With Framingham Cardiovascular Risk Score calculated for non-diseased individuals(men ≥15 and women ≥18 are classified as high cardiovascular risk).
  4. Perform an electrocardiogram for diagnose of arrhythmia.
  5. ABI, TBI, and baPWV are utilized to assess arteriosclerosis in the extremities, ABI < 0.9 or TBI < 0.7 or baPWV > 1400 cm/s is diagnostic of peripheral arterial disease.
  6. Carotid ultrasonography is performed to assess carotid plaque.
Prevalence of cognitive function | At 8-17 years postpartum
  Inquire about history of cognitive function(definitively diagnosed by a qualified physician).
Prevalence of renal disease | At 8-17 years postpartum
  Subjects who meet criterion 1 or 2 will be considered to have renal disease:
  1. Serum creatinine>133μmol/L.
  2. Urinary microalbumin/urinary creatinine>30mg/g.

SECONDARY OUTCOMES:
Prevalence of anxiety | At 8-17 years postpartum
  Assessed by standardized depression and anxiety scales [Zung Self-rating Anxiety Scale(SAS)].
  Anxiety Severity Classification:
  Normal: <50, Mild Anxiety: 50-59, Moderate Anxiety: 60-69, Severe Anxiety: ≥70
Thyroid Function | At 8-17 years postpartum
  Assessed via measurement of thyroid hormone levels
Bone Density | At 8-17 years postpartum
  Assessed via quantitative ultrasound (QUS) measurement of T-scores and Z-scores at the bilateral distal radius.
Offspring Growth and Development | At 8-17 years old
  Growth curve values persistently below the 3rd percentile (P3) or above the 97th percentile (P97), as defined by the *China Height and Weight Percentile Curves for Children and Adolescents Aged 2-18 Years* developed by the Growth and Development Research Laboratory, Capital Institute of Pediatrics, were considered indicative of abnormal growth
CAIDE Dementia Risk Score | At 8-17 years postpartum
  With CAIDE Dementia Risk Score calculated for individuals without history of cognitive function.
N-acetyl-β-D-glucosaminidase (NAG) | At 8-17 years postpartum
  >12U/L is considered early-stage renal tubule injury.
Prevalence of depression | At 8-17 years postpartum
  Assessed by standardized depression and anxiety scales [Zung Self-Rating Depression Scale(SDS)].
  Depression Severity Classification: Normal: <53, Mild Depression: 53-62, Moderate Depression: 63-72, Severe Depression: ≥73
Hyperuricemia | At 8-17 years postpartum
  Serum uric acid levels exceed 420 μmol/L.
Hyperhomocysteinemia | At 8-17 years postpartum
  Serum homocysteine >15 μmol/L
Fatty liver disease | At 8-17 years postpartum
  Liver Transient Elastography (CAP) Fat Attenuation Grading:
  Normal: <244 dB/m Mild Hepatic Steatosis: 244-269 dB/m Moderate Hepatic Steatosis: 269-296 dB/m Severe Hepatic Steatosis: >296 dB/m
Body fat percentage: | At 8-17 years postpartum
  18%-28% is considered normal.
Kutcher Adolescent Depression Scale (11-item version, KADS-11) | 11-17 years old
  Range: 0-33; Higher scores indicate worse status. A total score ≥9 suggests a depressive state.
Swanson, Nolan, and Pelham Rating Scale (SNAP-IV) | 10-18 years old
  Items 1-9 constitute the Attention Deficit subscale (range: 0-27, ≤13: Normal); Items 10-18 constitute the Hyperactivity-Impulsivity subscale (range: 0-27, ≤13: Normal); Items 19-26 constitute the Oppositional Defiant subscale: Abnormality is defined as ≥4 items scored as 2 or 3.
Screen for Child Anxiety Related Emotional Disorders (SCARED) | 10-18 years old
  Range: 0-82; Higher scores indicate worse condition; a total score ≥25 suggests anxiety.
Social Anxiety Scale for Children (SASC) | 10-18 years old
  Range: 0-20; Higher scores indicate worse condition; no standardized cutoff.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The clinical information of the participants and the primary outcome data of the LEGEND study will be shared
Supporting Information: Study Protocol, CSR
Time Frame: IPD will be available half year after the last participants finished the study